CLINICAL TRIAL: NCT01354548
Title: Prophylactic Training for the Prevention of Radiotherapy-induced Trismus - a Randomised Study. Health-related Quality of Life up to One Year After Radiotherapy in Patients With Head and Neck Cancer
Brief Title: Prevention of Trismus During Radiotherapy and Quality of Life in Head and Neck Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Linkoeping (Other)
Collaborators: Linkoeping University (Other Government); Ryhov County Hospital (Other)
Responsible Party: Principal Investigator, Vera Loorents, Project leader, University Hospital, Linkoeping
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FORSS-88571; The Swedish Cancer Society (Other Grant/Funding Number: The Swedish Cancer Society/CAN2009/1165); FoU (Other Grant/Funding Number: The medical research council of southeast sweden)
Record Dates: First submitted 2011-05-02; First posted 2011-05-17 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Trismus
Keywords: Trismus; Cancer; Radiotherapy; Quality of life
MeSH Terms: conditions — Trismus; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TheraBite grupp (Experimental)
  Interventions: Device: TheraBite® Jaw Motion Rehabilitation System™
- Conventional treatment (No Intervention)

INTERVENTIONS:
Device: TheraBite® Jaw Motion Rehabilitation System™ — A portable device which utilizes passive motion and stretching to improve mobility and flexibility of the jaw muscles and associated joints. Patients are given written and verbal information about TheraBite before the commencement of Radiotherapy. Investigators instruct on usage and maintenance of TheraBite. Patients are instructed to start a trainings pass by softening the jaw muscles with a simple exercise. The training programme consists of five stretches performed 5 times per day, each stretch held for 15 seconds, training continually during Radiation Therapy and up to one year after completion of Radiation Therapy.
  Arms: TheraBite grupp

SUMMARY:
Trismus (limited jaw mobility), can occur in patients undergoing radiotherapy to specific areas of the head or neck. Trismus leads to difficulty in eating, swallowing, speech and general mouth hygiene, which all have negative effects on quality of life. Research in the area of trismus is limited; it is not known exactly when trismus develops, one study suggests that some patients have experienced a diminished opening at as low doses as 15 Gy. Literature suggests benefits of a training programme, but there is a lack of evidence to support the use of a training programme during radiotherapy.

The purpose of this study is to investigate the effectiveness of a training programme during and after radiotherapy, and report the incidence of trismus in patients who receive radiotherapy to the jaw muscles. The study also investigates quality of life during radiotherapy and up to one year after completed treatment.

Patients who meet the criteria and give their consensus to the study are divided into two groups:

Group 1: Training with TheraBite Jaw Motion Rehabilitation System, which is a portable system utilizing repetitive passive motion and stretching to restore mobility and flexibility of the jaw musculature. Individuals train five times a day.

Group 2: Conventional treatment (jaw measurements once a week). If the individuals jaw mobility decreases 15% from the original start measurement, the patient is automatically offered a trainings program (as in group 1).

During radiation therapy a hospital specialist dentist measures the jaw mobility once a week, thereafter at 3,6,12 months after completed Radiation Therapy. On 5 different occasions the patients are requested to complete a Quality of life questionnaire. Patient's record their training frequency in a log book.

DETAILED DESCRIPTION:
Summary of the study programme

Background

During Radiation therapy to the mouth, throat or trachea can fibrosis often occur in the chewing muscles round the jaw causing a development of trismus (a limited jaw mobility). Trismus can cause pain, difficulty in eating, swallowing, speech and difficulty with general mouth hygiene. Despite the fact that this condition has been documented in older literature, there is limited research in the incidence of trismus. There is need of randomised studies to investigate the prevention of trismus both under and during Radiation Therapy.

Aims

The specific aims of this study are to investigate the effectiveness of Prophylactic training with a muscle warm-up programme and a mechanical device (TheraBite) to prevent trismus during Radiation Therapy and one year after completed therapy. The study also aims to investigate the incidence of radiotherapy-induced trismus in patients who receive radiotherapy to the masseter, temporalis, pterygoid muscles. Finally the study investigates whether trismus affects quality of life.

Methods

Patients

Sixty consecutive patients, from two different radiation clinics in Sweden, are randomised into the two different groups using a computer programme.

Treatment procedures

1. Intervention group: Daily training with a programme for TheraBite that trains passive movement, preceded by a warm-up programme. Mouth opening measurements are made once a week during treatment at the end of radiotherapy,three, six and 12 months after treatment.
2. Control group: Receiving traditional radiation therapy with nursing care, measuring the patients mouth opening once a week during treatment, at the end of radiation therapy,three, six, and 12 months after treatment. The same training programme as group one is offered to this group as soon as evidence of trismus develops.

This training is recorded by the patient in a log book. Weight, height, Mucositis analysis and quality of life are made before the commencement of radiation therapy, at the end of radiation therapy, three, six, and 12 months after treatment. The patient's weight is measured every week.

Results

The results of this study will give new and vital information that can give a basis to develop a clinical method of identifying and treating cancer patients who suffer from trismus. Thus giving new knowledge which can be used to formulate clinical practices.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Be able to communicate and understand the Swedish language.
* Compliance with training programme and follow-up during the study time period.
* Planed radiotherapy dose of at least 15Gy to the jaw muscles.
* Tooth 11 and 41 intact.

Exclusion Criteria:

* An operation in the target area that has already affected jaw mobility.
* Jaw measurement under 35mm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-02; Primary Completion 2016-04 (Actual); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Change in Jaw mobility measurement during Radiotherapy | Up to 7 weeks
  Proportion of participants free from trismus at the end of Radiotherapy.

SECONDARY OUTCOMES:
Change in Jaw Mobility measurement at 6 and 12 months after completed Radiotherapy | 6 and 12 months
  Proportion of participants free from trismus 6 and 12 months after completed Radiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Sussanne Börjeson, Med dr, Principal Investigator — Department of Medicine and Care, Division of Nursing Sciences, Faculty of Health Sciences, Linköping University, Sweden
Locations (2):
- Sweden (2):
  - Department of Radiation Oncology, Ryhov ,Sweden, Jönköping
  - Department of Radiation Oncology, University Hospital, Linkoping, Linköping

REFERENCES:
- See also: Link to the Medical research council of Southeast Sweden — http://www.fou.nu/is/forss/
- See also: Link to the Swedish cancer Society — http://www.cancerfonden.se/sv/Information-in-English/